CLINICAL TRIAL: NCT06634095
Title: The Effect of Using Moulage-Assisted Standardized Patient Simulation on Nursing Students
Brief Title: Effect of Moulage on Self-efficacy and Clinical Practice in Pressure Sores
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Fahri AŞKAN, Assistant Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024 03-04
Record Dates: First submitted 2024-09-14; First posted 2024-10-09 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Pressure Ulcers
Keywords: self-sufficiency; Moulage; Clinical Practice Regarding
MeSH Terms: conditions — Pressure Ulcer | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Experimental, randomised controlled, single-blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moulage group (Experimental): "It will consist of students trained with standardized patient simulation supported by a model."
  Interventions: Behavioral: Moulage group
- Contol group (No Intervention): Students in the control group will receive standard care.

INTERVENTIONS:
Behavioral: Moulage group — The experimental group is trained with a moulage-supported standardized patient simulation. Participants in the experimental group practice during the specified moulage-supported standardized patient simulation. Moulage-supported simulations regarding pressure ulcers will be created and training will be provided.
  Other Names: Control Group
  Arms: Moulage group

SUMMARY:
In the process of preventing, treating and caring for pressure ulcers, nurses take on an important responsibility and are one of the most common adverse events during hospitalizations worldwide. Pressure ulcers, which are a serious problem especially in cases requiring long-term care. These ulcers occur as a result of prolonged exposure of soft tissues to pressure and can lead to local tissue damage, carrying the risk of infection. In Turkey, pressure ulcers are considered an indicator of patient care quality for healthcare institutions, and many healthcare institutions continue their efforts to reduce the rate of pressure ulcers.

DETAILED DESCRIPTION:
Moulage-supported education provides appropriate care that increases the quality of care. Therefore, it is critical for nurses to develop pressure injury assessment skills before and after graduation. However, in clinical settings, there are challenges such as limited opportunities for developing psychomotor skills, increasing student numbers, complexity of the healthcare system, and patient safety issues. In response to these challenges, the importance of simulation-based education that provides practices similar to clinical experience has emerged. Moulage plays an important role in high-quality simulations that appeal to many senses. Moulage can be defined as the application of make-up or other elements to add realism to simulation training by creating realistic-looking wounds. The use of moulage provides a valuable opportunity for practical experience that can be perceived by many senses such as vision, hearing and touch. The use of moulage helps students understand the etiology, physiology and healing processes of the wound and is an effective tool for developing wound assessment skills.

Simulated patients, known as standardized patients, which have recently emerged, are used to promote performance, competence and knowledge development among nursing students. Standardized patients help students improve their clinical and speaking performances by providing them with the opportunity to realistically play the role of a patient with a health problem.

Evaluating nursing students' perceptions and thoughts about clinical practice and their self-efficacy perceptions can contribute to the development of more effective strategies by evaluating the effectiveness of clinical practice strategies.

No research has been found on the effect of the use of moulage-supported standardized patient simulation on nursing students' self-efficacy and clinical practice attitudes towards pressure ulcers. This study is planned to be conducted as an experimental study to investigate the effect of the use of moulage-supported standardized patient simulation on nursing students' self-efficacy and clinical practice attitudes towards pressure ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Students who have clinical field experience (internship),
* Volunteer to participate in the study,
* Have no attendance problems will be included in the study.

Exclusion Criteria:

* Students without clinical internship experience,
* Those who do not voluntarily participate in the work,
* Those with attendance issues will not be included in the work.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Pressure Injury Management Self-Efficacy Scale for Nurses | Baseline and 12 week
  Each item in the 10-item survey is scored from 1 (not competent at all) to 5 (completely competent). It should be measured using 0-100 points. The total score range to be obtained from the scale is 0-100.

SECONDARY OUTCOMES:
Attitude Scale for Nursing Students Towards Clinical Practices | Baseline and 12 week
  The scale items are of 5-point Likert type, scored as "Strongly disagree (1 point)", "Disagree (2 points)", "Undecided (3 points)", "Agree (4 points)" and Strongly Agree (5 points)". The lowest score that can be obtained from the scale is 26, the highest score is 130, and an increase in the total score indicates that students have developed a positive attitude towards clinical practice.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Van Yuzuncu Yıl University, Van, Tuşba
  - VAN YYU Faculty of Health Sciences, Van

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Celik H, Ozer M, Zincir H. Modification and Validation of the Vaccine Hesitancy Scale for Turkish Adult Vaccination. J Nurs Meas. 2024 Mar 14;32(1):82-94. doi: 10.1891/JNM-2022-0020. PMID 37827583
- [Result] Gilkey MB, McRee AL, Magnus BE, Reiter PL, Dempsey AF, Brewer NT. Vaccination Confidence and Parental Refusal/Delay of Early Childhood Vaccines. PLoS One. 2016 Jul 8;11(7):e0159087. doi: 10.1371/journal.pone.0159087. eCollection 2016. PMID 27391098
- [Result] Franklin MD, Schlundt DG, Wallston KA. Development and validation of a religious health fatalism measure for the African-American faith community. J Health Psychol. 2008 Apr;13(3):323-35. doi: 10.1177/1359105307088137. PMID 18420767
- [Result] Costa JC, Weber AM, Darmstadt GL, Abdalla S, Victora CG. Religious affiliation and immunization coverage in 15 countries in Sub-Saharan Africa. Vaccine. 2020 Jan 29;38(5):1160-1169. doi: 10.1016/j.vaccine.2019.11.024. Epub 2019 Nov 30. PMID 31791811
- [Result] Ahmed A, Lee KS, Bukhsh A, Al-Worafi YM, Sarker MMR, Ming LC, Khan TM. Outbreak of vaccine-preventable diseases in Muslim majority countries. J Infect Public Health. 2018 Mar-Apr;11(2):153-155. doi: 10.1016/j.jiph.2017.09.007. Epub 2017 Oct 4. PMID 28988775
- [Derived] Sarpdagi Y, Kaplan E, Sir O, Askan F, Yildiz M. The effect of moulage supported standardised patient simulation on nursing students' self-efficacy and clinical practice attitudes towards pressure injuries : A randomised controlled study. Nurse Educ Pract. 2026 Jan;90:104695. doi: 10.1016/j.nepr.2025.104695. Epub 2025 Dec 17. PMID 41420980